CLINICAL TRIAL: NCT07079657
Title: Thulium Laser and Growth Factors for Androgenetic Alopecia - a Prospective, Clinical Study
Brief Title: Thulium Laser and Growth Factors for Androgenetic Alopecia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Lynhda Nguyen, Dr. med., Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-23
Record Dates: First submitted 2025-07-13; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Androgenetic Alopecia (AGA)
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Thulium laser + growth factor serum + LED (Active Comparator): Thulium laser + growth factor serum + LED
  Interventions: Procedure: Thulium laser + growth factor serum + LED
- Thulium laser + growth factor serum (Active Comparator): Thulium laser + growth factor serum
  Interventions: Procedure: Thulium laser + growth factor serum
- Thulium laser (Active Comparator): Thulium laser
  Interventions: Procedure: Thulium laser

INTERVENTIONS:
Procedure: Thulium laser + growth factor serum + LED — 3 sessions at intervals of 6 weeks
  Arms: Thulium laser + growth factor serum + LED
Procedure: Thulium laser + growth factor serum — 3 sessions at intervals of 6 weeks
  Arms: Thulium laser + growth factor serum
Procedure: Thulium laser — 3 sessions at intervals of 6 weeks
  Arms: Thulium laser

SUMMARY:
Androgenetic alopecia (AGA) is a common cause of hair loss worldwide. It mainly affects the frontal and parietal regions of the scalp in up to 70 % of men and 40 % of women and has a significant negative psychological and emotional impact on those affected.

Various therapies are currently approved for the treatment of AGA in men and women, including topical minoxidil, topical or systemic finasteride, platelet-rich plasma and hair transplantation. In addition to these pharmacological and surgical interventions, laser therapies including thulium laser with growth factors have gained popularity.

Despite the clinical use of the thulium laser with growth factors in combination with LED phototherapy, there are only a few studies to date that have adequately investigated the objective and patient-side benefits of this therapy.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 and over
* Good general health, no relevant previous illnesses
* Presence of an AGA
* Cognitive ability and willingness to give consent (informed consent)
* Be willing and able to attend follow-up visits

Exclusion Criteria:

* Age < 18 years
* Pregnant or breastfeeding women
* Scarring alopecia, alopecia due to dermatoses (e.g. lichen ruber, lupus erythemodes,...), alopecia due to chemical or physical noxae, and other non-AGAs
* Significant scarring of the region to be treated
* Significant open wounds or lesions in the region to be treated
* Metallic implants in the head region
* Mental illnesses (psychoses, body perception disorders)
* Use of isotretinoin or other retinoids, psychotropic drugs, coumarins or heparins in the last 2 weeks
* Resurfacing (fractional, ablative, non-ablative) of the affected region < 2 months before and during the study period
* Tendency to excessive scarring
* Lack of informed consent and/or data protection declarations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Subject Global Aesthetic Improvement Scale | 1 and 6 months post-treatment
  scale from 0 (very much improved) to 4 (worse)
Hair density | at baseline, and 1 and 6 months post-treatment
  measurement of hair density before and after treatment
hair thickness | at baseline, and 1 and 6 months post-treatment
  hair thickness before and after treatment

SECONDARY OUTCOMES:
pain intensity | Periprocedural
  pain intensity during treatment using a numeric rating scale from 0 (no pain) to 10 (unbearable pain)

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Hamburg, Germany